CLINICAL TRIAL: NCT06389773
Title: Fostering Teamwork for Resilient Staff and Safe Care: Driving Post-pandemic Recovery and Renewal in Intensive Care Units
Brief Title: Teamwork for Resilient Staff and Safe Care in ICU
Acronym: FEARLESS_ICU
Status: Not yet recruiting | Type: Observational
Sponsor: King's College London (Other)
Responsible Party: Sponsor
Other Study IDs: 302958
Record Dates: First submitted 2024-04-25; First posted 2024-04-29 (Actual); Last update posted 2024-04-29 (Actual); Status verified 2024-04

CONDITIONS: Teamwork
Keywords: wellbeing; intensive care; patient safety

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this ethnographic study is to observe how healthcare professionals work together in an intensive care unit (ICU). The main questions it aims to answer are

* How do healthcare staff work together in everyday ICU settings?
* What helps people work together in ICUs?
* What challenges do staff face in working together in ICUs?
* How have teamwork practices changed since the COVID-19 pandemic?

Researchers will shadow staff during their day-to-day work. Key staff members will also be interviewed about their perceptions and experiences of teamwork.

DETAILED DESCRIPTION:
Teamwork impacts staff wellbeing and patient outcomes. This study focuses on the factors that facilitate or challenge teamworking practices in ICUs. A rapid ethnographic approach, including observation and interviews, ensures that what people say they do and what they actually do match up in practice. This project has two interrelated components: observation and one-on-one interviews.

Observations: A researcher will shadow various healthcare professionals in 10 different ICU units. These observations will cover multiple professions and different shift patterns, including handovers, ward rounds, and multi-disciplinary team meetings. This allows for a range of interactions to be covered which will elucidate how healthcare professionals work together. Written consent will be obtained from each healthcare professional shadowed, and researchers will observe in 20-minute blocks where possible to minimize burden. Researchers will record their observations in the form of fieldnotes which will be either hand-written or recorded on a dedicated iPad. Fieldnotes will later be expanded on, typed up, and pseudonymized. During this observation period, researchers may engage in informal discussions with healthcare professionals to clarify what they observe where appropriate though these will not be audio recorded. Additionally, while patients and their family members will provide verbal consent where possible for the researcher to be present in the room or at the bedside, data will not be collected on them.

All three members of the research team will visit each site; however, one researcher will remain at the site for the duration of the research period. Each site will incur a minimum of 75 observation hours over the course of four weeks.

Interviews: To supplement the observations, researchers will conduct one-on-one semi-structured interviews with key healthcare professionals in each study site. Initially, these individuals will be identified and approached by the researcher during the observation phase. Researchers will then employ a snowball method to identify further potential healthcare professionals to include. At least 15 healthcare professionals per site will be interviewed for this study. All healthcare professionals will provide their written consent for the interview.

Data analysis: All formal interview audio recordings will be recorded using a Dictaphone voice recorder with the participant's consent. These recordings will be transcribed using a King's College London approved transcription service and anonymised. Thematic analysis will be conducted to identify recurring themes (Braun and Clarke, 2006). The transcripts will be read and reread for familiarization before coding the data. During the coding process, a code book will be created with a list of codes and descriptions to accompany. To validate the coding, each researcher will code a small, random selection of the transcripts using the code book. Coding will be discussed to reach an agreement. Field notes obtained through observation will be spoken aloud by the researcher using a Dictaphone voice recorder and sent to the transcription service. The transcripts will be anonymized and uploaded to NVivo to be thematically analysed. The analysis will focus on answering the research questions, using constructs from the conceptual frameworks to sensitize the analysis.

ELIGIBILITY:
Inclusion Criteria:

* healthcare professionals
* work in an intensive care unit
* work in a selected case study site

Exclusion Criteria:

* not a healthcare professional (e.g. patients and their families)
* not working in an intensive care unit
* not working in a selected case study site

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: healthcare professionals working in a selected intensive care unit
Sampling Method: Non-Probability Sample
Enrollment: 75 (Estimated)
Dates: Start 2024-09-02 (Estimated); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Examine the changing nature of teamwork in ICUs in the post-pandemic context | 12 months
  Ethnographic data, including observational notes and interview transcripts will be collected and analysed using thematic analysis.

IPD SHARING:
Plan to Share IPD: No
Due to the ethnographic nature of the data collection, it will not be possible to make individual participant data available to other researchers.

REFERENCES:
- [Background] Xyrichis A, Rose L. Interprofessional collaboration in the intensive care unit: Power sharing is key (but are we up to it?). Intensive Crit Care Nurs. 2024 Feb;80:103536. doi: 10.1016/j.iccn.2023.103536. Epub 2023 Sep 30. No abstract available. PMID 37783179